CLINICAL TRIAL: NCT07038226
Title: Fecal Microbiota Transplantation Via Oral Capsule for Treating Refractory Constipation in Parkinson's Disease: a Double-blind, Placebo-controlled, Randomised Trial
Brief Title: Fecal Microbiota Transplantation Via Oral Capsule for Treating Refractory Constipation in Parkinson's Disease
Acronym: FORT-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyung Hee University Hospital (Other)
Collaborators: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Tae-Beom Ahn, Professor, Kyung Hee University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KHUH 2023-03-002-008; 2022 (Other Grant/Funding Number: CN Research Foundation)
Record Dates: First submitted 2025-06-04; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Constipation
Keywords: fecal transplantation; oral capsule
MeSH Terms: conditions — Parkinson Disease; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Block randomization is performed by an unblinded Clinical Research Associate (CRA), assigning participants to either the treatment group or the placebo group in a 1:1 ratio. All other researchers involved in the study remain blinded to group assignments. The researcher responsible for randomization does not engage in any other aspects of the research process. Randomization records are maintained separately from other clinical data to ensure confidentiality. Researchers, aside from the one handling randomization, are unaware of which participants are in the treatment or placebo group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive a visually identical capsule containing skim milk powder.
  Interventions: Biological: Placebo
- Oral capsule-delivered FMT (Experimental): Participants will receive oral capsules of lysophilized fecal microbiota.
  Interventions: Biological: Oral capsule-delivered FMT

INTERVENTIONS:
Biological: Placebo — a visually identical capsule containing skim milk powder
  Arms: Placebo
Biological: Oral capsule-delivered FMT — Oral capsules of lysophilized fecal microbiota
  Arms: Oral capsule-delivered FMT

SUMMARY:
The aim of this clinical trial is to assess the impact of fecal microbiota transplantation (FMT) delivered via oral capsules in patients with Parkinson's disease who suffer from refractory constipation. The primary questions this trial seeks to answer are:

Does FMT delivered through oral capsules improve constipation? Does FMT delivered through oral capsules enhance the motor symptoms associated with Parkinson's disease? Is FMT delivered through oral capsules safe for individuals with Parkinson's disease? Researchers will compare the intervention group with a control group to determine the presence of a placebo effect.

Participants in the study will:

Take antibiotics as a pre-treatment regimen for 5 days, followed by oral capsules containing either fecal microbiota or a placebo for 14 days.

Attend clinic visits at screening, visit 1 (baseline), visit 2 (4 weeks), and visit 3 (12 weeks).

Collect fecal samples and maintain a 2-week diary of their bowel habits before visits 1, 2, and 3.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 80 years.
* Voluntarily signed the informed consent form for participation in this study.
* Diagnosed with Parkinson's disease according to the UK Brain Bank Criteria.
* Either do not have or have controlled Parkinson's disease motor complications, allowing for stable use of anti-Parkinson's medication during the study period (12 weeks).
* Meet the definition of refractory constipation as follows:

A. On at least 1 out of 4 bowel movements, two or more of the following apply: i. Excessive straining.

ii. Lumpy/hard stools (Bristol Stool Form Scale 1-2). iii. Sensation of incomplete evacuation after defecation. iv. Sensation of anorectal obstruction or blockage. v. Manual maneuvers to facilitate defecation. vi. Fewer than three spontaneous bowel movements per week. B. Rarely experience loose stools without the use of laxatives. C. Symptoms began at least 6 months prior to diagnosis and have persisted for the past 3 months.

D. Constipation shows no improvement despite the use of various types of laxatives (bulk-forming, osmotic, saline, stimulant, or others) individually or in combination for at least 4 weeks.

Exclusion Criteria:

* Individuals with cognitive impairment scoring less than 20 on the Korean version of the Mini-Mental State Examination (K-MMSE).
* Individuals who have contraindications for fecal microbiota transplantation (acute infections, immunocompromised status, or a history of food allergies).
* Individuals with ileus or colonic pseudo-obstruction.
* Individuals with a history of major gastrointestinal surgeries, such as resection.
* Individuals with suspected or confirmed gastrointestinal obstruction or gastric outlet obstruction.
* Individuals with suspected or confirmed active gastrointestinal bleeding.
* Individuals with gastrointestinal diseases requiring treatment or medical consultation.
* Individuals receiving parenteral nutrition or enteral feeding.
* Individuals experiencing dysphagia symptoms (difficulty swallowing, choking during meals, etc.).
* Individuals who have taken antibiotics within 3 months prior to screening.
* Individuals who have participated in other drug clinical trials within 3 months prior to screening.
* Pregnant individuals.
* Individuals with other severe diseases that may impair quality of life or the ability to perform daily activities.
* Individuals with contraindications to the use of antibiotics (Ciprofloxacin, Metronidazole) as referenced in the text.
* Any other case where the researcher deems participation in the clinical trial to be inappropriate for the subject.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 39-Item Parkinson's Disease Questionnaire | Baseline up to Week 12
  The minimum score is 0 and the maximum score is 100, with higher scores indicating worse quality of life.
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | up to 12 weeks
  Any adverse effects derived from the intervention

SECONDARY OUTCOMES:
Change from baseline in Wexner Constipation Score | Baseline up to Week 12
  The minimum score is 0 and a maximum score is 30, with higher scores indicating more severe constipation.
Change from baseline in Bristol stool scale | Baseline up to Week 12
  The Bristol Stool Chart classifies stool types on a scale of 1 to 7, with 1 being the hardest and 7 being the most liquid.
Change from baseline in Geriatric Depression Scale-15 (short version) | Baseline up to Week 12
  The total score range is 0 to 15, with higher scores indicating more severe depressive symptoms.
Change from baseline in MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) with Hoehn and Yahr Stage (HYS) | Baseline up to Week 12
  The MDS-UPDRS has a total possible score of 260, with higher scores indicating greater disability. The HYS ranges from 0 to 5, or a clinical staging system that describes the progression of motor symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided